CLINICAL TRIAL: NCT07254000
Title: Anakinra Pilot 2 - A Study to Optimise Dose and Route of Administration of Anakinra in Preterm Infants
Acronym: AP2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Monash Medical Centre (Other)
Collaborators: Monash University (Other); Hudson Institute of Medical Research (Unknown); Liggins Institute (Other); Starship Children's Hospital of New Zealand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RES 24-0000-885A
Record Dates: First submitted 2025-04-07; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Premature Infants; Very Premature Infants; Inflammation
Keywords: anakinra; bronchopulmonary dysplasia; diffuse white matter injury; very premature infants
MeSH Terms: conditions — Premature Birth; Inflammation; Bronchopulmonary Dysplasia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: AP2 is a randomised, three-arm, parallel-group, dose-ranging trial to determine safety, efficacy and optimal dosing of intravenous anakinra in premature neonates, with subcutaneous pharmacokinetic sub-study. Neonates will be randomly assigned to 1 of 3 dosing levels (8 per group), with half of each dosing level assigned to recieve subcutaneous dosing in week 3.
  Population pharmacokinetic and physiology-based pharmacokinetic modelling will be employed to build on pharmacokinetic analysis from AP1, including multiple dose levels and subcutaneous dosing. Pooling of pharmacokinetic data from AP1 and AP2 (total n = 48) will enable establishment of a pharmacokinetic model, including key pharmacokinetic parameters clearance (CL), volume of distribution (VD), and absorption rate (Ka, subcutaneous) with sufficient precision (based on relative standard error) and model performance. In addition, PK will be linked through modelling with biomarkers and outcomes in expoloratory PKPD analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Anakinra dose 1 IV (Active Comparator): Anakinra IV for 21 days
  Interventions: Drug: Anakinra (Kineret®)
- Anakinra dose 1 IV/SC (Active Comparator): Anakinra IV for 14 days & SC for 7 days
  Interventions: Drug: Anakinra (Kineret®)
- Anakinra dose 2 IV (Active Comparator): Anakinra IV for 21 days
  Interventions: Drug: Anakinra (Kineret®)
- Anakinra dose 2 IV/SC (Active Comparator): Anakinra IV for 14 days & SC for 7 days
  Interventions: Drug: Anakinra (Kineret®)
- Anakinra dose 3 IV (Active Comparator): Anakinra IV for 21 days
  Interventions: Drug: Anakinra (Kineret®)
- Anakinra dose 3 IV/SC (Active Comparator): Anakinra IV for 14 days & SC for 7 days
  Interventions: Drug: Anakinra (Kineret®)

INTERVENTIONS:
Drug: Anakinra (Kineret®) — Standard care plus Anakinra for 21 days

SUMMARY:
A phase 2 randomised, three-arm, parallel-group, dose-ranging trial to determine safety, efficacy and optimal dosing of intravenous anakinra in premature neonates, with subcutaneous pharmacokinetic sub-study.

DETAILED DESCRIPTION:
Advances in neonatal intensive care have significantly improved the survival rates for extremely premature neonates. Despite this, many survivors develop chronic conditions such as cerebral palsy and chronic lung disease, primarily due to the pro-inflammatory environment common in these patients. Efforts to reduce these conditions using anti-inflammatory glucocorticoids are effective but are hindered by significant adverse effects that outweigh potential benefits for most neonates.

Crucially, not only is inflammation an important driver of morbidities of prematurity, but as shown by the investigators and other research groups, the potent pro-inflammatory cytokine interleukin-1 is a key player.

A phase I/IIa trial of anakinra in extremely premature infants (24 - 27+6 weeks gestational age) demonstrated feasibility of administration intravenous over the first 3 weeks of life, without any acute safety concerns and confirmation of mechanistic pharmacokinetic predictions.

The aims of this phase II dose-ranging trial (Anakinra Pilot 2, AP2) are to:

1. Establish pharmacokinetics, linearity and target concentration attainment over a range of doses, to determine optimal dosing regimen.
2. Assess feasibility and pharmacokinetics of an alternative route of administration (RoA), namely subcutaneous, in week 3 of treatment.
3. Further expand safety & feasibility, as well as perform exploratory pharmacometric dose-exposure-response analysis, against biomarkers and early efficacy endpoints.

The primary outcome is to refine understanding of anakinra population pharmacokinetics in extremely premature neonates, and at 3 different dosing levels, to allow determination of optimal dose for population target concentration attainment in future trials.

In addition, the pharmacokinetics of subcutaneously administered anakinra in extremely premature neonates (from week 3) will be explored. Population pharmacokinetic model development and validation, for intravenous and subcutaneous anakinra in premature neonates over the first 3 weeks of life, to enable dose determination for target concentration attainment.

Model performance and validation will be based on metrics and graphics of model 'goodness-of-fit', precision of parameter estimates (relative standard error & confidence intervals for CL, Vd and Ka) and predictive performance and robustness, per published (PMID: 27884052) and regulatory guidance (FDA guidance on Population Pharmacokinetics (https://www.fda.gov/regulatory-information/search-fda-guidance-documents/population-pharmacokinetics).

Population Pharmacokinetic (PK)/Pharmacodynamic (PD) Modeling will also enable exploratory investigation of the relationship between anakinra dose, concentration-time course in blood, and drug effects, both biomarkers of inflammation and clinical endpoints.

AP2 will recruit 24 infants born 24-28 weeks-GA, randomised to one of 3 dosing arms, 8 infants/arm, stratified to ensure balanced GA-distribution. Participants will otherwise receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Born between 24+0 and 28+6 weeks of gestation

Exclusion Criteria:

* Inability of the legal representatives to consent,
* Genetic syndromes,
* Severe cardiac anomalies,
* Substantial pre-/perinatal compromise,
* Congenital diaphragmatic hernia,
* Intrauterine stroke,
* Conditions that could confound trial results
* Imminent death or plan for comfort / palliative care
* Infants born outside the recruiting institutions

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Population Pharmacokinetics (PopPK) Model of the Clearance of anakinra in extremely premature neonates from birth, during the 3-week treatment period. | From Baseline up to Day 21
  Point Estimate of Population Total Clearance (CL) of anakinra will be reported.
Population Pharmacokinetics (PopPK) Model of the Volume of Distribution of anakinra in extremely premature neonates from birth, during the 3-week treatment period. | From Baseline up to Day 21
  Point Estimate of Population Volume of Distribution (VD) of anakinra will be reported.
Population Pharmacokinetics (PopPK) Model of the Absorption of Population of subcutaneously administered anakinra in extremely premature neonates from birth, during the 3-week treatment period. | Day 14-21
  Point Estimate of Population Absorption of subcutaneously administered anakinra will be reported.

SECONDARY OUTCOMES:
Incidence of bronchopulmonary dysplasia | 4 months.
  Early efficacy endpoints (exploratory): incidence of bronchopulmonary dysplasia, in comparison to contemporary unit and national statistics.
Hammersmith infant neurological examination | 6 months
  Early efficacy endpoint (exploratory): Hammersmith infant neurological examination; performed at 3-4 months of corrected age, in comparison to contemporary unit and national statistics.
Incidence of intracranial/intraventricular haemorrhage and peri-ventricular leukomalacia. | 4 months
  Early efficacy endpoint (exploratory): incidence of intracranial/intraventricular haemorrhage and peri-ventricular leukomalacia, in comparison to contemporary unit and national statistics.
Safety of anakinra in extremely premature neonates. | 4 weeks
  Safety of anakinra IV and SC in premature neonates, at 3 dosing levels, measured as incidence of safety endpoints in particular late-onset sepsis and necrotizing enterocolitis (compared with contemporary unit and national statistics) as well as neutropenia, thrombocytopenia, acute kidney injury, drug-induced liver injury (per Hy's Law).
Individual Total Clearance (CL) of anakinra in extremely premature neonates. | From Baseline up to Day 21.
  Average of individual model-derived estimates of CL will be reported.
Individual Volume of Distribution (VD) of anakinra in extremely premature neonates. | Baseline to Day 21.
  Average of individual model-derived estimates of VD will be reported.
Individual Absorption Rate Constant (Ka) of subcutaneously administered anakinra in extremely premature neonates. | Day 14-21.
  Average of individual model-derived estimates of Ka will be reported.
Individual Maximum Serum Concentration (Cmax) of anakinra. | Baseline to Day 21.
  Average of individual model-derived estimates of Cmax will be reported.
Individual Area Under the Concentration-time Curve Within a Dosing Interval (AUCtau) of anakinra. | Baseline to D21.
  Average of individual model-derived estimates of AUCtau will be reported.
Individual Model - derived Ctrough Concentrations of anakinra. | Baseline to D21.
  Average of individual model-derived Ctrough concentrations of anakinra will be reported.

OTHER OUTCOMES:
Feasibility of 3 weeks of anakinra administration to extremely premature neonates from birth, both intravenously and subcutaneously. | 1 month
  Feasibility of anakinra IV and SC in premature neonates, at 3 dosing levels, measured as succesful completion of intervention treatment course, including subcutaneous dosing.
Influence of anakinra on microbiome. | 3 weeks
  Monitoring for lung and gut microbiome changes during the treatment course by collection and analysis of bronchoalveolar lavage fluid (in intubated infants), nasopharyngeal swabs, and stool.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Model of the Effect of anakinra Systemic Exposure on clinical endpoints. | 4 months
  Point Estimate of population IC50 of anakinra associated with a reduction in incidence of early efficacy endpoints (exploratory), including bronchopulmonary dysplasia, intracranial/intraventricular haemorrhage & peri-ventricular leukomalacia, and Hammersmith infant neurological examination; performed at 3-4 months of corrected age.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Model of the Effect of anakinra Systemic Exposure on biomarkers of the inflammatory cascade. | 4 Months.
  Point Estimate of population IC50 of anakinra, i.e. the drug concentration required to produce 50% of maximal inhibition of the IL-1-driven inflammatory cascade. Biomarkers investigated will include cellular proteomic biomarkers of inflammatory activity and inhibition, including lymphoid and myeloid cell polarisation and activation as well as responsiveness to stimulants such as lipopolysaccharide (LPS) and PMA/ionomycin during the treatment course.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Model of the Effect of anakinra Systemic Exposure on adverse effects. | Baseline to Day 21.
  Point Estimate of population EC50 of anakinra, i.e. the drug concentration associated with exploratory safety endpoints including late-onset sepsis, necrotizing enterocolitis, neutropenia, thrombocytopenia, acute kidney injury, drug-induced liver injury (per Hy's Law).

CONTACTS AND LOCATIONS:
Overall Officials: Marcel F Nold, Prof, Principal Investigator — Monash Health/ Monash University/ Hudson Institute of Medical Research; Claudia Nold, Prof, Principal Investigator — Hudson Institute of Medical Research; Rod Hunt, Prof, Principal Investigator — Monash Health / Monash University; Robert Galinsky, Dr, Principal Investigator — Hudson Institute of Medical Research; Gergely Toldi, Dr, Principal Investigator — Starship Children's Hospital / Liggins Institute; Carl Kirkpatrick, Prof, Principal Investigator — Monash University; David Metz, Dr, Principal Investigator — Monash Health / Royal Children's Hospital
Locations (2):
- Monash Children's Hospital, Clayton, Victoria, Australia
- Starship Children's Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No